CLINICAL TRIAL: NCT00837226
Title: The Effects of Weight Loss From Bariatric Surgery on Intraocular Pressure
Brief Title: Effects of Weight Loss From Bariatric Surgery on Intraocular Pressure (IOP)
Acronym: IOP
Status: Withdrawn | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Robert Feldman, ◦Clinical Professor and Chair and Richard S. Ruiz, M.D., Distinguished University Chair in Ophthalmology, The University of Texas Health Science Center, Houston
Other Study IDs: 08-0499
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study group-Bariatric procedure performed
- Control group: No bariatric procedures

SUMMARY:
The purpose of this study is to determine if there is an effect on the eye pressure from extreme weight loss by bariatric procedures. The hypothesis is that excess fat in the orbit of the eye compresses on the outflow system, which causes an elevated eye pressure. This can have many consequences, including the risk for glaucoma. We hope to establish if there is an effect between eye pressure and weight.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Written informed consent obtained
* BMI > 40 kg/m2 without associated comorbidities or > 35 kg/m2 with associated comorbidities. In the normal indication for routine bariatric surgery, comorbidities include hypertension, type II diabetes, venous stasis, sleep apnea, polycystic ovary syndrome, pseudotumor cerebri, nonalcoholic steatohepatitis, gastroesophageal reflux disease, coronary artery disease, degenerative joint disease, cancer, and hypercholesterolemia.

Exclusion Criteria:

* Current use of systemic steroids
* Any systemic medication which is unstable and can affect IOP
* History or evidence of glaucoma
* Any ocular trauma or ocular surgery
* Outside normal range of corneal thickness (500-600 microns)
* Unable to follow-up for 3 years
* Participating in any investigational device or medication study within 30 days of baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are included in this study will have been evaluated for bariatric surgery and will meet the current eligibility requirements for bariatric surgery. These requirements include that the patient must have failed dietary therapy and have a BMI(body mass index) greater than 40 kg/m2 without associated comorbidities or have a BMI greater than 35 kg/m2 with associated comorbidities. Eleven subjects who will be evaluated for bariatric surgery but choose not to undergo the surgery will be recruited to serve as controls and to verify the changes in intraocular pressure (IOP) are due to the weight loss. It is expected that the IOP of the control patients will be relatively stable, assuming the patients will not have any other surgery or intervention which could affect the IOP.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | Data will be recorded the same day when a patient comes to the clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Feldman, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Minimally Invasive Surgeons of Texas, Bellaire, Texas, United States